CLINICAL TRIAL: NCT06158737
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial Evaluated the Safety and Tolerability, Pharmacokinetic and Pharmacodynamics Profile, and Immunogenicity of a Single Dose of JS010 Injection in Healthy Subjects
Brief Title: A Clinical Trial Evaluated the Safety and Tolerability, Pharmacokinetic and Pharmacodynamics Profile, and Immunogenicity of a Single Dose of JS010 Injection in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: JS010-001
Record Dates: First submitted 2023-11-07; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: JS010 injection (Experimental)
  Interventions: Drug: JS010 injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS010 injection — This study adopts a dose escalation design with six preset dose levels, namely 3mg, 30mg, 150mg, 300mg,600mg, 900mg, single subcutaneous injection. A total of 48 healthy subjects were enrolled in the experiment, 8 in each group.They were randomly assigned to receive JS010 injection and matching placebo in a ratio of 3:1. In accordance with the dose-escalation principle,Starting from the lowest initial dose, increasing to the higher dose and proceeding in sequence. Each subject can receive only one dose Level of single subcutaneous administration.
  Arms: Experimental: JS010 injection
Drug: Placebo — This study adopts a dose escalation design with six preset dose levels, namely 3mg, 30mg, 150mg, 300mg,600mg, 900mg, single subcutaneous injection. A total of 48 healthy subjects were enrolled in the experiment, 8 in each group.They were randomly assigned to receive JS010 injection and matching placebo in a ratio of 3:1. In accordance with the dose-escalation principle,Starting from the lowest initial dose, increasing to the higher dose and proceeding in sequence. Each subject can receive only one dose Level of single subcutaneous administration.
  Arms: Placebo

SUMMARY:
This study adopts a dose escalation design with six preset dose levels, namely 3mg, 30mg, 150mg, 300mg,600mg, 900mg, single subcutaneous injection. A total of 48 healthy subjects will be enrolled in the experiment, 8 in each group.They will be randomly assigned to receive JS010 injection and matching placebo in a ratio of 3:1. In accordance with the dose-escalation principle,Starting from the lowest initial dose, increasing to the higher dose and proceeding in sequence. Each subject can receive only one dose Level of single subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands and voluntarily signs a written informed consent form (ICF).
* Healthy male or female subjects aged 18-45 years (inclusive) at the time of signing informed consent.
* The body mass index (BMI) at screening was in the range of 18.5~28.0kg/m2 (inclusive).
* Female subjects must meet the following conditions: no fertility (e.g. documented hysterectomy, bilateral transfusion;

Blood pregnancy detection knot during ovular tubule resection or ligation, or menopause for more than 1 year), or screening of fertile persons' results were negative, and they were willing to use strict and effective contraceptive methods (such as medication or barrier methods) during the study period.

Male subjects were required to consent to a strict and effective form of contraception.

· Subjects are willing and able to complete the procedures and examinations associated with the trial, and can maintain a stable diet, exercise and ohter lifestyle habits during the trial.

Exclusion Criteria:

* Subjects' forearm skin could not be stimulated by capsaicin, or was unresponsive or abnormally responsive to capsaicin stimulation.
* There is medical history or clinical evidence that the subject has a serious acute or chronic illness (including, but not limited to:

Heart, kidney, nerve, endocrine, blood, immune, infection, metabolic dysfunction, etc.), by investigator judged that participating in the study could confound the results or put the subjects at risk.

* There is obvious concomitant disease, or physical examination, laboratory examination, chest X-ray, abdominal B-ultrasound, and electrocardiogram which reveals any clinically significant abnormalities, discomfort or disease. According to the researchers, it is not in line with clinical practice.
* There is a history of malignancy, except for carcinoma in situ that has been completely resected surgically.
* Drug abuse or alcohol dependence within the last 1 year.
* A known history of HIV and/or syphilis infection, or a positive test for HIV and/or syphilis antibodies at screening;
* Known history of hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection, or hepatitis B surface at the time of screening

Antigen (HBsAg) and/or hepatitis C antibody positive.

* Had undergone abdominal surgery or endoscopic intestinal surgery within 6 months prior to randomization.
* Had undergone major surgical treatment within 6 months prior to randomization.
* Had received hospitalization within 3 months prior to randomization.
* Blood donation or blood loss ≥300ml in the 3 months prior to randomization.[17] Previously received drugs that target CGRP or CGRP receptors.
* Use of any therapeutic or investigational biologics in the 6 months prior to randomization.
* Participated in any of the trial drug interventions within 3 months or 5 half-lives (whichever is older) prior to randomization

The clinical study.

· Had used any prescription drugs or drugs within 30 days prior to randomization or 5 half-lives, whichever is older

Remedies, including Chinese herbs, vitamins and dietary supplements (hormones used in contraception for women of childbearing age)

Except for birth control pills).

* Received live vaccine within 30 days prior to randomization.
* A history of allergy to biological agents, including monoclonal antibodies.
* A history of severe allergies to food, drugs, insect bites, etc.
* Pregnant and lactating women.
* Any other situation in which the investigator deems it inappropriate to participate in the study, such as the subject having potential compliance problems; Unable to complete all inspections and evaluations as required by the programme

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-09-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 168 days post-dose
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) , as well as abnormalities in vital signs, electrocardiogram and laboratory tests.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 168 days post-dose
  Peak Plasma Concentration of JS010
Time to Maximum Plasma Concentration (Tmax) | up to 168 days post-dose
  Time to Maximum Plasma Concentration of JS010
Terminal Elimination Half-Life (t1/2) | up to 168 days post-dose
  Terminal Elimination Half-Life (t1/2) of JS010
Area Under the Plasma Concentration Versus Time Curve (AUC) | up to 168 days post-dose
  Area Under the Plasma Concentration Versus Time Curve of JS010
Cutaneous blood flow | up to 168 days post-dose
  The rate of change in cutaneous blood flow at each time point was calculated and descriptive statistics were performed
Anti-drug antibodies (ADA) | up to 168 days post-dose
  JS010 Incidence and titer of anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No